CLINICAL TRIAL: NCT01260961
Title: Developing Treatment, Treatment Validation and Treatment Scope in the Setting of an Autism Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sherie Novotny, M.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0220080189
Record Dates: First submitted 2010-11-23; First posted 2010-12-15 (Estimated); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docosa Hexanoic Acid (Active Comparator)
  Interventions: Dietary Supplement: Docosahexanoic Acid
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — The volunteers will start on the 200 mg daily of the placebo and will not increase their dose during the study.
  Arms: Placebo
Dietary Supplement: Docosahexanoic Acid — The volunteers will start on the 200 mg daily of the DHA capsule and will not increase their dose during the study.
  Other Names: DHA
  Arms: Docosa Hexanoic Acid

SUMMARY:
Dr. Sherie Novotny of the Department of Psychiatry at UMDNJ-RWJMS and collaborators are starting a treatment trial to determine whether Docosa Hexanoic Acid(DHA), the major omega-3 fatty acid found in the brain and a component of fish oil, has any effects on the symptoms of autism.

We propose to carry out a trial to test the effect of DHA compared to a placebo (a pill with no drug in it) on several aspects of autism in children and adolescents, in a 12-week clinical study with children or adolescents in the age group of 5-17 with a diagnosis of Autism Spectrum Disorder. Additionally this trial will study genes related to the therapeutic agent, DHA, and biomarkers related to DHA in the urine.

DETAILED DESCRIPTION:
Growing evidence supports oxidative stress may contribute to autism. Docosa Hexanoic Acid(DHA)is a normal substance that is present in large amounts in the brain and can be used by the body to produce natural antioxidants. Our hope is that supplementing DHA in individuals with autism may improve some aspects of their functioning. Specifically our aims are:

Aim 1. To assess the effect of DHA vs. placebo treatment on the global severity of child and adolescent autistic disorder, via a 12-week double blind placebo-controlled parallel study. Global severity will be assessed by the Autism Diagnostic Observation Schedule-Generic (ADOS-G) and additionally in younger children by the Vineland Adaptive Behavior Scale.

Aim 2. To assess the effect of DHA vs. placebo treatment on behavioral symptoms and functional ability in children with autism. Assessment will be by the Aberrant Behavior Checklist (ABC)-Community Version11.

Aim 3. To develop an improved protocol and study design based upon these studies for future large scale studies of DHA in the autistic population.

Aim 4. Monitor the effects of therapy on the isoprostane biomarker. Aim 5: Develop additional biomarkers that correlate with autism and with therapy. We will extend the analyses to neuroprostanes and resolvins. We will measure: (i) Urinary excretion of the isoprostane metabolites, 2,3 Dinor-5,6 dihydro-PGF2t and iPF4α-VI. (ii) DHA derived resolvins D2, D4, D5 and D6 and neuroprotectin.

Aim 6: Confirm our preliminary results by correlating increased isoprostane excretion with GSTM1*0 copy number in individuals with autism.

Aim 7: In the same way, correlate GSTM1*0 copy number with response to therapy assessed by diminution of isoprostane excretion during therapy.

Aim 8: Study additional biomarkers developed through Hypothesis #2 for correlation with GSTM1*0 copy number and response to therapy to identify additional gene-biomarker correlations.

Aim 9: Study additional polymorphisms of genes related to DHA metabolism, for association with autism, gene-biomarker correlations, and correlation with response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV, ADI, and ADOS criteria for autistic disorder
* Age 5-17.
* Outpatients
* Parent or legal guardian signing informed consent, and assent documented for patient with demonstrated capacity to provide it.
* Sexually active females of childbearing potential must use an acceptable method of birth control (oral contraceptive medications [the administration of which must be supervised by a parent or guardian], IUD, depot medication, double barrier or tubal ligation) and have a negative serum pregnancy test prior to entry into the study.
* Subjects with history of seizures, who have been seizure-free for more than or equal to 6 months on a stable dose of anticonvulsant medication.Non-medicated subjects with a history of seizures who have been seizure-free for more than or equal to 6 months.Subjects with abnormal EEG but no clinical seizures.

Exclusion Criteria:

* Subjects who are pregnant or nursing mothers.
* Sexually active females of childbearing potential who are not using adequate birth control measures (detailed above in inclusion criteria).
* Subjects with overall adaptive behavior scores below the age of two years on the Vineland Adaptive Behavior Rating Scale.
* Subjects with active or unstable epilepsy.
* Subjects with any of the following past or present mental disorders: schizophrenia, schizoaffective disorder, major depressive disorder, bipolar I or II disorders or substance abuse disorders.
* Subjects who are a serious suicidal risk.
* Subjects with clinically significant or unstable medical illness that would contraindicate participation in the study, including hematopoietic or cardiovascular disease, pancreatitis, liver toxicity, and polycystic ovary syndrome
* Subjects reporting history of encephalitis, phenylketonuria, tuberous sclerosis, fragile X syndrome, anoxia during birth, pica, neurofibromatosis, hypomelanosis of Ito, hypothyroidism, Duchenne muscular dystrophy, and maternal rubella.
* Patients with history of the following:gastrointestinal, liver, or kidney, or other known conditions which will presently interfere presently with the absorption, distribution, metabolism, or excretion of drugs, cerebrovascular disease or brain trauma, clinically significant unstable endocrine disorder, such as hypo- or hyperthyroidism, recent history or presence of any form of malignancy
* Treatment within the previous 30 days with any drug known to a well-defined potential for toxicity to a major organ
* Subjects with clinically significant abnormalities in laboratory tests or physical exam
* Subjects likely to require ECT.
* Subjects unable to tolerate taper from psychoactive medication if necessary.
* Subjects with a history of hypersensitivity or severe side effects associated with the use of divalproex sodium, or other an ineffective prior therapeutic trial of omega three fatty acids.
* Subjects who have received any of the following interventions within the prescribed period before starting treatment-investigational drugs within the previous 30 days.
* Subjects who have begun any new alternative non-medication treatments, such as diet, vitamins, and psychosocial therapy, within the previous three months.
* Subjects with any organic or systemic disease or patients who require a therapeutic intervention, not otherwise specified, which would confound the evaluation of the safety of the study medication.
* Subjects who reside in a remote geographical area who do not have regular access to transportation to the clinical facility.
* If a patient is not doing well enough (defined by CGI-AD Severity score of 3-"mildly ill" or better)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2010-11; Primary Completion 2015-07 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Amelioration of phenotypic features of autism | three years
  Amelioration of phenotypic features of autism as measured by a significant decrease from the baseline, in global severity of autism score and Aberrant Behavior Checklist scores

SECONDARY OUTCOMES:
oxidative stress biomarkers | Three years
  We will be measuring isoprostane 8-iso-PGF2a.
  The measurements will be in ng mg Creatinine and we expect a significant decrease in levels from the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sherie Novotny, MD, Principal Investigator — Rutgers-RWJMS
Locations (1):
- Rutgers, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No